CLINICAL TRIAL: NCT05704686
Title: Visual Outcomes and Patient Satisfaction After the Implantation of Isopure Extended-Depth-of-Focus Intraocular Lens (EDOF-IOL), With a Mini-Monovision Target
Brief Title: Clinical Outcomes of an New EDOF IOL (Isopure®)
Status: Completed | Type: Observational
Sponsor: Kristof Vandekerckhove, MD, MBA (Other)
Responsible Party: Sponsor-Investigator, Kristof Vandekerckhove, MD, MBA, Medical Director and Founder, Vista Alpina Eye Clinic, Vista Alpina Eye Clinic
Organization: Vista Alpina Eye Clinic (Other)
Other Study IDs: Iso123
Record Dates: First submitted 2023-01-19; First posted 2023-01-30 (Actual); Last update posted 2023-01-30 (Actual); Status verified 2023-01

CONDITIONS: Lens Opacities; Cataract; Pseudophakia
MeSH Terms: conditions — Cataract; Pseudophakia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Isopure 1.2.3 intraocular EDOF lens implantation — Bilateral Isopure 1.2.3 intraocular EDOF IOL implantation during a routine cataract surgery.

SUMMARY:
Single-center, retrospective, open-label observational study aiming to evaluate visual outcomes and patient satisfaction after bilateral implantation of Isopure® EDOF-IOL with a mono-minovision target.

DETAILED DESCRIPTION:
This single-center retrospective study investigates visual outcomes and patient satisfaction in subjects bilaterally implanted with Enhanced-Depth of Focus (EDOF) Isopure® IOL during routine bilateral cataract surgery.

The study is carried out in an ophthalmic clinic in Switzerland. In this study, routine surgical techniques and postoperative follow-up will be applied as for all other (non-study) cataract patients in the clinic. Therefore, all study patients will be operated in immediate consecutive bilateral mode (routine in clinic). Patients participating in this study will be recruited and enrolled postoperatively. They undergo routine postoperative follow-up examinations, and data are collected at the third scheduled examination (4 to 6 weeks after surgery) and at a telephone call 4 to 6 months after surgery.

Isopure 1.2.3 is a CE certified intraocular lens readily available on the market in Switzerland.

The primary outcome consists in demonstrating a preserved distance visual acuity while improving binocular spectacle-free intermediate vision and, to a lesser extent, near vision. Binocular defocus curves are measured for each participant to simulate visual acuity at different distances. Patient satisfaction with treatment and subjective ratings of visual phenomena will be assessed using a modified PRISQ questionnaire and a modified NEI quality of vision questionnaire (RQL-42) at the third postoperative visit and three months after surgery.

At Vista Alpina Eye Clinic, mini-monovision is routinely used to further improve binocular intermediate and near vision while preserving the quality of distance vision in patients implanted bilaterally with EDOF Isopure® IOLs. Analysis of the retrospective data should help support this surgical strategy.

Patients with astigmatism up to 1.5 D benefit intraoperatively from Opposite Clear Corneal Incisions (OCCI) to reduce astigmatism. Analysis of our retrospective data will allow comparison of their visual performance with that of patients without astigmatism who did not require an additional OCCI procedure.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients aged 50 years or older undergoing a routine cataract surgery and benefiting from bilateral IOL implantation with Isopure 1.2.3 IOL;
* Patient's willingness to participate in the study;
* Capacity to understand and sign an informed consent form and comply with examination procedures;
* Cataractous eyes with no vision-impacting comorbidity (estimated visual potential post-surgery 0.2 logMAR or better);
* Regular total corneal astigmatism ≤1.5 D (measured by topography method)

Exclusion Criteria:

* Cooperation difficulties (distance from home, general health conditions, cognitive impairment);
* Subjects with diagnosed extra- or intraocular vision-affecting comorbidities (macular degeneration, glaucoma or other retinal or optic nerve disorders, previous ocular surgeries, amblyopia);
* Patients who previously benefitted from refractive surgery (PRK/LASIK) were included if no refractive surgery-related complications were noted (i.e: ectasia, corneal haze, dry eye);
* History or presence of macular edema;
* Perioperative complications;
* Congenital, uveitic, traumatic or surgically-complicated cataract
* Regular total corneal astigmatism >1.5 dioptres (measured by topography method)
* Irregular cornea, including keratotomy

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consecutive patients undergoing routine cataract surgery and having opted for the implantation of an EDOF intraocular lens, in a primary ophthalmic clinic in Switzerland.
Sampling Method: Probability Sample
Enrollment: 62 (Actual)
Dates: Start 2021-04-26 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
UDVA(m) | 4-6 weeks postoperatively
  Monocular Uncorrected Distance Visual Acuity
CDVA(m) | 4-6 weeks postoperatively
  Monocular Corrected Distance Visual Acuity
UDVA(b) | 4-6 weeks postoperatively
  Binocular Uncorrected Distance Visual Acuity
UIVA | 4-6 weeks postoperatively
  Binocular Uncorrected Intermediate Visual Acuity (80 cm)
UNVA | 4-6 weeks postoperatively
  Binocular Uncorrected Near Visual Acuity (40 cm)
Defocus curve | 4-6 weeks postoperatively
  Binocular distance-corrected defocus curve analysis simulating visual acuities at different distances.

SECONDARY OUTCOMES:
Patient satisfaction with the visual outcome | 4-6 weeks postoperatively and 4-6 months postoperatively
  (modified) PRISQ questionnaire
Subjective rating of visual phenomena | 4-6 weeks postoperatively and 4-6 months postoperatively
  (modified) NEI quality of vision questionnaire (RQL-42, questions 17 and 38)

OTHER OUTCOMES:
Impact of OCCI on residual refractive cylinder | 4-6 weeks postoperatively
  Residual refractive cylinder in eyes undergoing OCCI (eyes with preoperative topographic total corneal astigmatism 0.6 - 1.5 diopters), compared to eyes not having undergone OCCI (preoperative topographic cylinder 0 - 0.5 diopters).
Impact of OCCI on uncorrected binocular visual acuity | 4-6 weeks postoperatively
  Comparison of binocular UDVA between three subgroups. Subgroup 1: both eyes having undergone OCCI. Subgroup 2: one eyes having undergone OCCI. Subgroup 3: none of the eyes having undergone OCCI.
Impact of OCCI on uncorrected monocular visual acuity | 4-6 weeks postoperatively
  Comparison of monocular UDVA between eyes having undergone OCCI and eyes not having undergone OCCI (eyes with emmetropic objective only)
Accuracy of different IOL-formulas | 4-6 weeks postoperatively
  Comparing various IOL-formulas used to calculate the appropriate IOL power during preoperative assessment. The objective is to determine which IOL formulas are most accurate, overall, and (subgroups) in function of the anatomy of the eye (short vs long eyes, shallow versus deep anterior chamber)

CONTACTS AND LOCATIONS:
Overall Officials: Kristof Vandekerckhove, MD, Principal Investigator — Vista Alpina Eye Clinic
Locations (1):
- Vista Alpina Eye Clinic, Visp, Switzerland

IPD SHARING:
Plan to Share IPD: No